CLINICAL TRIAL: NCT00059306
Title: Secondary Prevention of Small Subcortical Strokes (SPS3) Trial
Brief Title: Secondary Prevention of Small Subcortical Strokes Trial
Acronym: SPS3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H09-03016; CRC
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Cerebrovascular Accident; Hypertension
Keywords: stroke; hypertension; high blood pressure; lacunar stroke; subcortical stroke; aspirin; clopidogrel
MeSH Terms: conditions — Stroke; Hypertension; Stroke, Lacunar | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiplatelet (Active Comparator): Participants receive aspirin + placebo OR aspirin + clopidogrel
  Interventions: Drug: aspirin; Drug: clopidogrel; Other: placebo
- Blood pressure (Active Comparator): The goal of the blood pressure aspect of this trial is to find out if lowering blood pressure after stroke helps to prevent recurrent stroke and preserves cognition.
  Interventions: Other: Target of Blood Pressure

INTERVENTIONS:
Drug: aspirin — Participants receive aspirin + placebo, specifically: aspirin (325 mg) with placebo (an inactive substance). Participants will take 1 of each pill a day until the end of the study.
  Arms: Antiplatelet
Drug: clopidogrel — Participants will receive aspirin + clopidogrel, specifically: aspirin (325 mg) with clopidogrel (75 mg)-- Participants will take 1 of each pill a day until the end of the study.
  Arms: Antiplatelet
Other: Target of Blood Pressure — Participants will be assigned to one of 2 groups of blood pressure control. The difference between the two groups is the target level of systolic blood pressure-either 130-149 mmHg or below 130 mmHg; to do so, the scientists will use medications that are already in the market for blood pressure management.
  Arms: Blood pressure
Other: placebo — an inactive substance
  Arms: Antiplatelet

SUMMARY:
The goal of this study is to learn if combination antiplatelet therapy (aspirin and clopidogrel) is more effective than aspirin alone for the prevention of recurrent stroke and cognitive decline, and if intensive blood pressure control is associated with fewer recurrent strokes and cognitive decline.

On July 21, 2011 the DSMB recommended terminating the anti platelet arm of the study due to an imbalance of overall and major non-CNS hemorrhagic SAE's and total deaths in the investigational anti platelet combination of aspirin + clopidogrel and an interim statistical analysis that demonstrated futility in the investigational anti platelet arm. It was recommended that patients be continued on standard care of aspirin mono therapy until their study close-out visit. Also, recommended the continuation and completion of the plood pressure arm following the protocol.

DETAILED DESCRIPTION:
Stroke is damage to the brain caused by problems in the blood vessels. Strokes often cause paralysis, loss of sensation and speech, and other problems. A lacunar or small Subcortical stroke affects the inner part of the brain causing small "pea sized" areas of damage due to blockage of small blood vessels within the brain.

This multi-center study will recruit 3000 participants (20 percent of whom will be Hispanic) to find out if using aspirin and clopidogrel is more effective than using aspirin alone to prevent recurrent stroke in patients with lacunar stroke confirmed by MRI, and if lowering a patient's blood pressure below the usual limits will also help prevent recurrent stroke and maintain thinking ability. Both aspirin and clopidogrel are widely-used for blood clotting and stroke prevention. Investigators intend to find out if using the drugs together is more effective than using aspirin alone.

Participants will be randomly assigned to one of 2 types of treatment: either aspirin alone or the combination of aspirin and clopidogrel. In addition, participants will be assigned to one of 2 groups of blood pressure control. The difference between the two groups is the target level of systolic blood pressure-either 130-149 or below 130. The goal of the blood pressure aspect of this trial is to find out if lowering blood pressure after stroke helps to prevent recurrent stroke and preserves cognition.

ELIGIBILITY:
INCLUSION:

Small subcortical ischemic stroke or subcortical TIA.

Inclusion criteria are based on TOAST criteria supplemented by required MRI data. All of the following criteria must be met:

* One of the lacunar stroke clinical syndromes (adapted from Fisher) lasting > 24 hrs within the past 6 months
* Absence of signs or symptoms of cortical dysfunction such as aphasia, apraxia, agnosia, agraphia, homonymous visual field defect, etc.
* No ipsilateral cervical carotid stenosis (≥50%) by a reliable imaging modality done in an approved laboratory since the qualifying small subcortical stroke (S3), if hemispheric.
* No major-risk cardioembolic sources requiring anticoagulation or other specific therapy. Minor-risk cardioembolic sources will be permitted if anticoagulation is not prescribed by the patient's primary care physician.
* Subcortical TIA with corresponding lesion on DWI.
* MRI evidence of S3: a. Presence of an S3 (1.5 and 2 cm in diameter corresponding to the qualifying event on DWI; when TIA, ADC image must confirm lesion or T2/FLAIR (hyperintense lesions) (required for all brainstem events) OR multiple S3s on FLAIR/TI(<1.5 cm in diameter) (hypointense lesions) b. Absence of cortical stroke and large subcortical stroke (recent or remote).

EXCLUSION:

To be eligible for entry into the study, the patient must not meet any of the criteria listed below:

* Disabling stroke (Modified Rankin Scale less than or equal to 4)
* Previous intracranial hemorrhage (excluding traumatic) or hemorrhagic stroke
* Age under 30 years
* High risk of bleeding (e.g. recurrent GI or GU bleeding, active peptic ulcer disease, etc)
* Anticipated requirement for long-term use of anticoagulants (e.g. recurrent DVT) or other antiplatelets
* Prior cortical stroke (diagnosed either clinically or by neuroimaging), or prior cortical or retinal TIA
* Prior ipsilateral carotid endarterectomy
* Impaired renal function: GFR <40
* Intolerance or contraindications to aspirin or clopidogrel (including thrombocytopenia, prolonged INR)
* A score < 24 (adjusted for age and education) on the Folstein Mini Mental Status Examination
* Medical contraindication to MRI
* Pregnancy or women of child-bearing potential who are not following an effective method of contraception
* Geographic or social factors making study participation impractical
* Unable or unwilling to provide informed consent
* Unlikely to be compliant with therapy/unwilling to return for frequent clinic visits
* Patients concurrently participating in another study with an investigational drug or device
* Other likely specific cause of stroke (e.g. dissection, vasculitis, prothrombotic diathesis, drug abuse)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3020 (Actual)
Dates: Start 2003-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically defined ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by non-investigational CT or MRI | Mean follow up of 4 years
Evidence of hemorrhagic stroke; a neurologic deficit associated with intraparenchymal or subarachnoid space lesion on CT/MRI or cerebral hemorrhage demonstrated by surgery or autopsy. | within mean follow-up of 4 years

SECONDARY OUTCOMES:
The difference in the rate of cognitive decline among SPS3 participants assigned to receive aspirin alone versus combination of aspirin and clopidogrel, assessed through repeated neuropsychological tests; and major vascular events. | within mean follow-up of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Benavente, M.D., Principal Investigator — University of British Columbia; Robert Hart, M.D., Principal Investigator — McMaster University
Locations (63):
- United States (39):
  - University of Southern Alabama Stroke Center, Mobile, Alabama
  - Catholic Healthcare West, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arizona, Department of Neurology, Tucson, Arizona
  - University of California San Diego Medical Center, San Diego, California
  - University of California San Francisco-Fresno, San Francisco-Fresno, California
  - Denver, Englewood, Colorado
  - Melbourne, Melbourne, Florida
  - Miami-University of Miami, Miller School of Medicine, Miami, Florida
  - Emory University, Grady Health System, Atlanta, Georgia
  - Mercy Medical Center-Ruan Neurology Clinical Research, Des Moines, Iowa
  - University of Kentucky, Aging/Stroke Program, Lexington, Kentucky
  - Suburban Hospital, Bethesda, Maryland
  - Boston University, Boston, Massachusetts
  - Wayne State, Detroit, Michigan
  - Henry Ford Hospital, Department of Neurology, Detroit, Michigan
  - Berman Center, Minneapolis, Minnesota
  - Mayo Stroke Center KA-SL-13, Rochester, Minnesota
  - University of Washington, Sant Louis, Missouri
  - Tenet Health, St. Louis University, St Louis, Missouri
  - St. John's Mercy, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Buffalo, Buffalo, New York
  - Helen Hayes Hospital, Haverstraw, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University, Sciences-Neurology, Winston-Salem, North Carolina
  - Case Western, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Ohio State University, Division of Stroke, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Scurlock Stroke Center, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Washington, Seattle, Washington
  - Marshfield Clinic, Department of Neurology, Marshfield, Wisconsin
  - Medical College of Wisconsin-Neurology, Milwaukee, Wisconsin
- Canada (8):
  - Calgary Health, Calgary, Alberta
  - SPS3 Coordinating Center, Vancouver, British Columbia
  - Halifax, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Greenfield Park, Greenfield Park, Quebec
  - McGill-Jewish General, Montreal, Quebec
  - McGill-Montreal General, Montreal, Quebec
  - CHA-Hospital de l'Enfant-Jesus, Québec, Quebec
- Chile (2):
  - Hospital Clinico de la Universidad Católica de Chile, Santiago
  - Hospital Naval Almirante Nef, 'Subida Alessandri s/n, Hall A, Oficina 9, Viña del Mar
- Hospital-Clinica Kennedy, Guayaquil, Ecuador
- Mexico (4):
  - Hospital de La Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León
  - Antiguo Hospital Civil de Guadalajara, Guadalajara
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zuibrán, Mexico City
  - Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez, Mexico City
- Hospital Sabogal Essalud-Unidad de Investigacion, Bellavista-Callao, Lima, Peru
- Spain (8):
  - Hosp. Universitario Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Passeig Marítim 25-29, Barcelona
  - Hospital de la Santa Creu I Sant Pau, c/Sant Antoni Maria Claret, 167, Barcelona
  - Hospital del Sagrat Cor. Quinta de Salut I'Alianca, c/Viladomat 288, Barcelona
  - Hosp. Parc Tauli de Sabadell, Barcelona
  - Hosp. de Girona Dr. Josep Trueta, Girona
  - Hospital La Paz, Madrid
  - Universidad de Santiago de Compostela, Facultad de Medicina y Odontologia, Santiago de Compostela

REFERENCES:
- [Derived] Goldstein ED, Liew SQR, Shu L, Yaghi S. The impact of pre-stroke aspirin exposure on radiographic appearance and disability outcomes: A post-hoc analysis of the SPS3 trial: Aspirin Use and Small Subcortical Stroke. J Stroke Cerebrovasc Dis. 2024 Mar;33(3):107566. doi: 10.1016/j.jstrokecerebrovasdis.2024.107566. Epub 2024 Jan 10. PMID 38214239
- [Derived] Anadani M, Turan TN, Yaghi S, Spiotta AM, Gory B, Sharma R, Sheth KN, de Havenon A. Change in Smoking Behavior and Outcome After Ischemic Stroke: Post-Hoc Analysis of the SPS3 Trial. Stroke. 2023 Apr;54(4):921-927. doi: 10.1161/STROKEAHA.121.038202. Epub 2023 Mar 6. PMID 36876480
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Shihab S, Boucher RE, Abraham N, Wei G, Beddhu S. Influence of Baseline Diastolic Blood Pressure on the Effects of Intensive Systolic Blood Pressure Lowering on the Risk of Stroke. Hypertension. 2022 Apr;79(4):785-793. doi: 10.1161/HYPERTENSIONAHA.121.18172. Epub 2022 Feb 4. PMID 35114798
- [Derived] Cukierman-Yaffe T, McClure LA, Risoli T, Bosch J, Sharma M, Gerstein HC, Benavente O. The Relationship Between Glucose Control and Cognitive Function in People With Diabetes After a Lacunar Stroke. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1521-e1528. doi: 10.1210/clinem/dgab022. PMID 33481011
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Blum MR, Scherzer R, Ikeme JC, Benavente OR, McClure LA, Peralta CA, Odden MC. Functional health and white matter hyperintensities as effect modifiers of blood pressure-lowering on cognitive function and vascular events in older Secondary Prevention of Small Subcortical Strokes trial participants. J Hypertens. 2020 Aug;38(8):1578-1585. doi: 10.1097/HJH.0000000000002440. PMID 32371759
- [Derived] Agarwal A, Cheung AK, Ma J, Cho M, Li M. Effect of Baseline Kidney Function on the Risk of Recurrent Stroke and on Effects of Intensive Blood Pressure Control in Patients With Previous Lacunar Stroke: A Post Hoc Analysis of the SPS3 Trial (Secondary Prevention of Small Subcortical Strokes). J Am Heart Assoc. 2019 Aug 20;8(16):e013098. doi: 10.1161/JAHA.119.013098. Epub 2019 Aug 19. PMID 31423869
- [Derived] Ikeme JC, Pergola PE, Scherzer R, Shlipak MG, Catanese L, McClure LA, Benavente OR, Peralta CA. Cerebral White Matter Hyperintensities, Kidney Function Decline, and Recurrent Stroke After Intensive Blood Pressure Lowering: Results From the Secondary Prevention of Small Subcortical Strokes ( SPS 3) Trial. J Am Heart Assoc. 2019 Feb 5;8(3):e010091. doi: 10.1161/JAHA.118.010091. PMID 30686103
- [Derived] Magvanjav O, McDonough CW, Gong Y, McClure LA, Talbert RL, Horenstein RB, Shuldiner AR, Benavente OR, Mitchell BD, Johnson JA; NINDS SiGN (Stroke Genetics Network). Pharmacogenetic Associations of beta1-Adrenergic Receptor Polymorphisms With Cardiovascular Outcomes in the SPS3 Trial (Secondary Prevention of Small Subcortical Strokes). Stroke. 2017 May;48(5):1337-1343. doi: 10.1161/STROKEAHA.116.015936. Epub 2017 Mar 28. PMID 28351962
- [Derived] Wilson LK, Pearce LA, Arauz A, Anderson DC, Tapia J, Bazan C, Benavente OR, Field TS; SPS3 Investigators. Morphological classification of penetrating artery pontine infarcts and association with risk factors and prognosis: The SPS3 trial. Int J Stroke. 2016 Jun;11(4):412-9. doi: 10.1177/1747493016637366. Epub 2016 Mar 8. PMID 26956031
- [Derived] Boehme AK, McClure LA, Zhang Y, Luna JM, Del Brutto OH, Benavente OR, Elkind MS. Inflammatory Markers and Outcomes After Lacunar Stroke: Levels of Inflammatory Markers in Treatment of Stroke Study. Stroke. 2016 Mar;47(3):659-67. doi: 10.1161/STROKEAHA.115.012166. PMID 26888535
- [Derived] Peralta CA, McClure LA, Scherzer R, Odden MC, White CL, Shlipak M, Benavente O, Pergola P. Effect of Intensive Versus Usual Blood Pressure Control on Kidney Function Among Individuals With Prior Lacunar Stroke: A Post Hoc Analysis of the Secondary Prevention of Small Subcortical Strokes (SPS3) Randomized Trial. Circulation. 2016 Feb 9;133(6):584-91. doi: 10.1161/CIRCULATIONAHA.115.019657. Epub 2016 Jan 13. PMID 26762524
- [Derived] Odden MC, McClure LA, Sawaya BP, White CL, Peralta CA, Field TS, Hart RG, Benavente OR, Pergola PE. Achieved Blood Pressure and Outcomes in the Secondary Prevention of Small Subcortical Strokes Trial. Hypertension. 2016 Jan;67(1):63-9. doi: 10.1161/HYPERTENSIONAHA.115.06480. Epub 2015 Nov 9. PMID 26553236
- [Derived] McDonough CW, McClure LA, Mitchell BD, Gong Y, Horenstein RB, Lewis JP, Field TS, Talbert RL, Benavente OR, Johnson JA, Shuldiner AR. CYP2C19 metabolizer status and clopidogrel efficacy in the Secondary Prevention of Small Subcortical Strokes (SPS3) study. J Am Heart Assoc. 2015 May 27;4(6):e001652. doi: 10.1161/JAHA.114.001652. PMID 26019129
- [Derived] Pearce LA, McClure LA, Anderson DC, Jacova C, Sharma M, Hart RG, Benavente OR; SPS3 Investigators. Effects of long-term blood pressure lowering and dual antiplatelet treatment on cognitive function in patients with recent lacunar stroke: a secondary analysis from the SPS3 randomised trial. Lancet Neurol. 2014 Dec;13(12):1177-85. doi: 10.1016/S1474-4422(14)70224-8. Epub 2014 Oct 23. PMID 25453457
- [Derived] Field TS, McClure LA, White CL, Pergola PE, Hart RG, Benavente OR, Hill MD; SPS3 Investigators. Should Blood Pressure Targets After Lacunar Stroke Vary by Body Size? The SPS3 Trial. Am J Hypertens. 2015 Jun;28(6):756-64. doi: 10.1093/ajh/hpu228. Epub 2014 Dec 1. PMID 25452300
- [Derived] Asdaghi N, Pearce LA, Nakajima M, Field TS, Bazan C, Cermeno F, McClure LA, Anderson DC, Hart RG, Benavente OR; SPS3 Investigators. Clinical correlates of infarct shape and volume in lacunar strokes: the Secondary Prevention of Small Subcortical Strokes trial. Stroke. 2014 Oct;45(10):2952-8. doi: 10.1161/STROKEAHA.114.005211. Epub 2014 Sep 4. PMID 25190442
- [Derived] Sharma M, Pearce LA, Benavente OR, Anderson DC, Connolly SJ, Palacio S, Coffey CS, Hart RG. Predictors of mortality in patients with lacunar stroke in the secondary prevention of small subcortical strokes trial. Stroke. 2014 Oct;45(10):2989-94. doi: 10.1161/STROKEAHA.114.005789. Epub 2014 Aug 26. PMID 25158772
- [Derived] Palacio S, McClure LA, Benavente OR, Bazan C 3rd, Pergola P, Hart RG. Lacunar strokes in patients with diabetes mellitus: risk factors, infarct location, and prognosis: the secondary prevention of small subcortical strokes study. Stroke. 2014 Sep;45(9):2689-94. doi: 10.1161/STROKEAHA.114.005018. Epub 2014 Jul 17. PMID 25034716
- [Derived] Benavente OR, Pearce LA, Bazan C, Roldan AM, Catanese L, Bhat Livezey VM, Vidal-Pergola G, McClure LA, Hart RG; SPS3 Investigators. Clinical-MRI correlations in a multiethnic cohort with recent lacunar stroke: the SPS3 trial. Int J Stroke. 2014 Dec;9(8):1057-64. doi: 10.1111/ijs.12282. Epub 2014 May 27. PMID 24862645
- [Derived] Lewis BL, Pearce LA, Field TS, White CL, Benavente OR; SPS3 Investigators. The relevance of living supports on antiplatelet adherence and trial participation: the SPS3 trial. Int J Stroke. 2014 Jun;9(4):443-8. doi: 10.1111/ijs.12267. Epub 2014 Mar 24. PMID 24661819
- [Derived] Elkind MS, Luna JM, McClure LA, Zhang Y, Coffey CS, Roldan A, Del Brutto OH, Pretell EJ, Pettigrew LC, Meyer BC, Tapia J, White C, Benavente OR; LIMITS Investigators. C-reactive protein as a prognostic marker after lacunar stroke: levels of inflammatory markers in the treatment of stroke study. Stroke. 2014 Mar;45(3):707-16. doi: 10.1161/STROKEAHA.113.004562. Epub 2014 Feb 12. PMID 24523037
- [Derived] Dhamoon MS, McClure LA, White CL, Lau H, Benavente O, Elkind MS. Quality of life after lacunar stroke: the Secondary Prevention of Small Subcortical Strokes study. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):1131-7. doi: 10.1016/j.jstrokecerebrovasdis.2013.09.029. Epub 2013 Oct 28. PMID 24177006
- [Derived] White CL, Pergola PE, Szychowski JM, Talbert R, Cervantes-Arriaga A, Clark HD, Del Brutto OH, Godoy IE, Hill MD, Pelegri A, Sussman CR, Taylor AA, Valdivia J, Anderson DC, Conwit R, Benavente OR; SPS3 Investigators. Blood pressure after recent stroke: baseline findings from the secondary prevention of small subcortical strokes trial. Am J Hypertens. 2013 Sep;26(9):1114-22. doi: 10.1093/ajh/hpt076. Epub 2013 Jun 4. PMID 23736109
- [Derived] SPS3 Study Group; Benavente OR, Coffey CS, Conwit R, Hart RG, McClure LA, Pearce LA, Pergola PE, Szychowski JM. Blood-pressure targets in patients with recent lacunar stroke: the SPS3 randomised trial. Lancet. 2013 Aug 10;382(9891):507-15. doi: 10.1016/S0140-6736(13)60852-1. Epub 2013 May 29. PMID 23726159
- [Derived] Jacova C, Pearce LA, Costello R, McClure LA, Holliday SL, Hart RG, Benavente OR. Cognitive impairment in lacunar strokes: the SPS3 trial. Ann Neurol. 2012 Sep;72(3):351-62. doi: 10.1002/ana.23733. PMID 23034910
- [Derived] SPS3 Investigators; Benavente OR, Hart RG, McClure LA, Szychowski JM, Coffey CS, Pearce LA. Effects of clopidogrel added to aspirin in patients with recent lacunar stroke. N Engl J Med. 2012 Aug 30;367(9):817-25. doi: 10.1056/NEJMoa1204133. PMID 22931315
- [Derived] Palacio S, Hart RG, Pearce LA, Benavente OR. Effect of addition of clopidogrel to aspirin on mortality: systematic review of randomized trials. Stroke. 2012 Aug;43(8):2157-62. doi: 10.1161/STROKEAHA.112.656173. PMID 22826359
- [Derived] McClure LA, Szychowski JM, Benavente O, Coffey CS. Sample size re-estimation in an on-going NIH-sponsored clinical trial: the secondary prevention of small subcortical strokes experience. Contemp Clin Trials. 2012 Sep;33(5):1088-93. doi: 10.1016/j.cct.2012.06.007. Epub 2012 Jun 30. PMID 22750086
- [Derived] Graves JW, White CL, Szychowski JM, Pergola PE, Benavente OR, Coffey CS, Hornung LN, Hart RG; SPS3 Study Investigators. Predictors of lowering SBP to assigned targets at 12 months in the Secondary Prevention of Small Subcortical Strokes study. J Hypertens. 2012 Jun;30(6):1233-40. doi: 10.1097/HJH.0b013e328353968d. PMID 22499292
- [Derived] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Derived] Benavente OR, White CL, Pearce L, Pergola P, Roldan A, Benavente MF, Coffey C, McClure LA, Szychowski JM, Conwit R, Heberling PA, Howard G, Bazan C, Vidal-Pergola G, Talbert R, Hart RG; SPS3 Investigators. The Secondary Prevention of Small Subcortical Strokes (SPS3) study. Int J Stroke. 2011 Apr;6(2):164-75. doi: 10.1111/j.1747-4949.2010.00573.x. Epub 2011 Jan 26. PMID 21371282
- [Derived] Elkind MS, Luna JM, Coffey CS, McClure LA, Liu KM, Spitalnik S, Paik MC, Roldan A, White C, Hart R, Benavente O. The Levels of Inflammatory Markers in the Treatment of Stroke study (LIMITS): inflammatory biomarkers as risk predictors after lacunar stroke. Int J Stroke. 2010 Apr;5(2):117-25. doi: 10.1111/j.1747-4949.2010.00420.x. PMID 20446946
- See also: Related Info — http://sps3.med.ubc.ca/
- See also: Related Info — http://www.nlm.nih.gov/databases/alerts/2011_ninds_stroke.html